CLINICAL TRIAL: NCT07232459
Title: Clinical Study of [18F]FT8 PET/CT in Evaluating Amyloidosis
Brief Title: [18F]FT8 PET Imaging in Immunoglobulin Light Chain Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University
Other Study IDs: TJMUGH-12
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Amyloid; Cardiac Amyloidosis; Amyloidosis; Healthy Subjects
Keywords: PET/CT; Cardiac amyloidosis; immunoglobulin light chain
MeSH Terms: conditions — Alzheimer Disease; Amyloid Neuropathies, Familial; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Participants will receive a single intravenous bolus injection of 10 ± 3 mCi of [18F]FT8 followed by a PET/CT scan.
  Interventions: Diagnostic Test: [18F]FT8
- Amyloidosis Patients: Participants will receive a single intravenous bolus injection of 10 ± 3 mCi of [18F]FT8, followed by a PET/CT scan.
  Interventions: Diagnostic Test: [18F]FT8

INTERVENTIONS:
Diagnostic Test: [18F]FT8 — Each subject will receive a single intravenous injection of [18F]FT8 and will undergo PET imaging at a specified time.

SUMMARY:
[18F]FT8, a derivative of 1-(4-pyridyl)-4-piperazinyl arene ([18F]TPZA), exhibits high affinity for AL amyloid in myocardial tissue sections and shows no significant binding to transthyretin amyloid. By comparing its diagnostic performance against established clinical methods, including echocardiography, contrast-enhanced MRI, and relevant laboratory tests, this study aims to establish [18F]FT8 as the basis for a robust PET protocol for the direct visualization and differential diagnosis of AL amyloidosis . The study preimarily evaluates the safety and diagnostic efficacy of [18F]FT8 PET imaging in human subjects.

DETAILED DESCRIPTION:
Subjects will undergo [18F]FT8 PET/CT scans for safety and diagnostic efficacy evaluation. Organ uptake will be quantified using the standard uptake value (SUV). Clinical assessments and laboratory tests, including baseline information collection, physical examination, cardiac function assessment, and hepatic and renal function tests, will be conducted before and after the scan.

ELIGIBILITY:
1. Subject Recruitment Participants will be recruited from outpatients and/or inpatient populations of the Hematology Department at Tianjin Medical University General Hospital. The principal investigator and collaborating hematologists will ensure consistent application of diagnosis and enrollment criteria based on standardized guidelines. The planned enrollment includes 20 patients with systemic amyloidosis (including cardiac involvement) and 5 healthy volunteers.
2. Amyloidosis Patients:

2.1 Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Adult patients (age ≥ 18 years);
2. Suspected, newly diagnosed, or previously diagnosed with cardiac amyloidosis, with supporting evidence from one or more of the following: cardiac MRI, contrast-enhanced CT, serum biomarkers (e.g., NT-proBNP, Troponin), or histopathological confirmation of amyloidosis.
3. Scheduled to undergo a clinical Pan-Amyloid PET/CT scan as part of standard care or clinical evaluation.
4. Able to understand the study procedures and provide written informed consent. 2.2 Exclusion Criteria

Subjects will be excluded based on any of the following:

1. Confirmed non-cardiac amyloidosis or other non-amyloid cardiac pathologies that could confound image interpretation.
2. Pregnancy or breastfeeding.
3. Any medical, psychological, or social condition that, in the opinion of the investigator, would compromise the subject's ability to participate fully or complete the study follow-up.

3. Healthy Volunteers: 3.1 Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Adult subjects (age ≥ 18 years);
2. No clinical evidence of active cardiac or systemic disease, as confirmed by medical history review, physical examination, and electrocardiogram (ECG).
3. Able to understand the study procedures and provide written informed consent. 3.2 Exclusion Criteria:

Subjects will be excluded based on any of the following:

1. History or current diagnosis of any significant cardiac, hepatic, renal, or neurological disorder.
2. Pregnancy or breastfeeding.
3. Any condition that, in the opinion of the investigator, could pose an increased risk from the study procedure or interfere with the interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with confirmed or suspected systemic or cardiac amyloidosis, including cases secondary to hematologic disorders or genetic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2028-07-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
The safety assessment | From time of injection up to 7 days post-injection
  The incidence of adverse events assessed by the investigator as related to the [18F]FT8 injection. Systematically collect and assess all adverse events within 7 days post-injection through physical examinations, vital signs monitoring, clinical laboratory tests (complete blood count, hepatic and renal function). All events will be graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
[18F]FT8 Organ Uptake measured by Standardized Uptake Value (SUV) | At the time of the single [18F]FT8 PET/CT scan (Day 1)
  Quantification of [18F]FT8 uptake in major organs (e.g., heart, liver, kidneys) using the Standardized Uptake Value (SUV). This measurement will be performed on the PET/CT scans acquired at a specified time. The outcome will be reported as the SUV for each organ in both amyloidosis patients and control subjects.

SECONDARY OUTCOMES:
The Biodistribution of [18F]FT8 in subjects | At the time of the single [18F]FT8 PET/CT scan (Day 1)
  Semi-quantitatively evaluate the tracer's uptake in the interest organs (including heart, liver, kidneys, lungs, brain, bones, thyroid, blood pool, and other related organs) by measuring the Standard Uptake Value (SUV).
Radiation Dosimetry | At the time of the single [18F]FT8 PET/CT scan (Day 1)
  Calculate the effective radiation dose (mSv) to various human organs and the whole body.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No